CLINICAL TRIAL: NCT04365582
Title: A Randomized Trial of Efficacy and Safety of an Early OUTpatient Treatment of COVID-19 in Patients With Risk Factor for Poor Outcome: a Strategy to Prevent Hospitalization
Brief Title: OUTpatient Treatment of COVID-19 in Patients With Risk Factor for Poor Outcome
Acronym: OUTCOV
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The PI decided.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUTCOV
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-04

CONDITIONS: COVID
Keywords: COVID; outpatient; ambulatory; prognosis
MeSH Terms: interventions — Azithromycin; Hydroxychloroquine; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Azithromycin (Experimental): Azithromycin
  Interventions: Drug: Azithromycin
- Hydroxychlororquine (Experimental): Hydroxychlororquine
  Interventions: Drug: Hydroxychloroquine
- Lopinavir/Ritonavir (Experimental): Lopinavir/Ritonavir
  Interventions: Drug: Lopinavir 200Mg/Ritonavir 50Mg Tab
- standards of care (No Intervention): SoC

INTERVENTIONS:
Drug: Azithromycin — 500 mg day 1 ; 250 mg/day for 4 days
  Arms: Azithromycin
Drug: Hydroxychloroquine — 200 mg x 3/day for 10 days
  Arms: Hydroxychlororquine
Drug: Lopinavir 200Mg/Ritonavir 50Mg Tab — 400/100 mg (2 tablets) x 2/day for 15 days
  Other Names: Lopinavir/Ritonavir
  Arms: Lopinavir/Ritonavir

SUMMARY:
COVID-19 is a respiratory disease due to a novel coronavirus (SARS-CoV-2) that causes substantial morbidity and mortality. To date, no treatment has been proved to be effective in COVID-19. Elderly patients and patients with comorbidities have the worse prognosis with a higher risk of hospitalization, ICU admission and death. The efficacy of an early outpatient treatment could be suggested but need to be confirmed. This confirmation is mandatory to improve prognosis of COVID-19 but also to avoid unsuspected deleterious effect of drugs already used in clinical practice but not based on evidence.

DETAILED DESCRIPTION:
The investigators make the hypothesis that an early outpatient treatment of COVID among patient with respiratory symptoms and risk factors for poor outcome can improve the prognosis of these patient and decrease the need for hospital admission.

Our study is an open label randomized clinical trial comparing 4 arms of treatment: Standards of Care (SoC) alone versus SoC + Azithromycine versus SoC + Hydroxychloroquine vs Soc + Lopinavir/Ritonavir.

Our involved population is patients more than 50 years of age with comorbidity or patients more than 70 years of age.

Our primary objective is to evaluate the efficacy of early outpatient treatment compared to standard of care in patients COVID-19 with risk factors for poor outcome. The criteria is hospital admission at Day 20 and the hospital admission rate will be compared between groups by a Chi² test or a Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

1. Either patients over 50 years of age with at least one comorbidity (hypertension, diabetes, obesity, cancer, chronic renal disease, immunodeficiency) OR patients over 70 years of age with or without comorbidity
2. Laboratory (PCR-) proved infection by COVID-19 or radiological sign highly suggestive of COVID-19
3. Respiratory symptoms (cough, chest discomfort, dyspnea)
4. Affiliation to the social security network
5. Able to understand and sign a written informed consent form

Exclusion Criteria:

1. Need for hospitalization according to updated French guidelines (ministère de la santé_04/04/2020)
2. Patient in long-term care facility
3. Patient without concern confirmation of COVID-19 by laboratory (PCR swab) test or chest CT
4. Known hypersensitivity or contra-indication to the 3 experimental treatments (azithromycin, hydroxychloroquine, lopinavir/ritonavir).
5. Any reason making follow up of the patient impossible during the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Hospital admission | Day 20
  Hospitalization at D20

SECONDARY OUTCOMES:
Effect of treatment on Death at D20 | Day 20
  This outcome corresponds to the number of patients who died on day 20.
Effect of treatment on Death at D60 | Day 60
  This outcome corresponds to the number of patients who died on day 60.
Effect of treatment on Death due to COVID at D20 | Day 20
  This outcome corresponds to the number of patients who died due to COVID on day 20.
Effect of treatment on Death due to COVID at D60 | Day 60
  This outcome corresponds to the number of patients who died due to COVID on day 60.
Effect of treatment on need for ICU stay at D20 | Day 20
  This outcome corresponds to the number of participants who need ICU stay at day 20.
Effect of treatment on need for ICU stay at D60 | Day 60
  This outcome corresponds to the number of participants who need ICU stay at day 60.
Effect of treatment on duration of ICU stay at D20 | Day 20
  This outcome evaluates the duration of patient's ICU stay at day 20.
Effect of treatment on duration of ICU stay at D60 | Day 60
  This outcome evaluates the duration of patient's ICU stay at day 60.
Effect of treatment on need of mechanical ventilation at D20 | Day 20
  This outcome corresponds to the number of participants who need mechanical ventilation at D20.
Effect of treatment on need of mechanical ventilation at D60 | Day 60
  This outcome corresponds to the number of participants who need mechanical ventilation at D60.
Effect of treatment on duration of mechanical ventilation at D20 | Day 20
  This outcome corresponds to the duration of patient's mechanical ventilation at D20.
Effect of treatment on duration of mechanical ventilation at D60 | Day 60
  This outcome corresponds to the duration of patient's mechanical ventilation at D60.
Effect of treatment on time to hospitalization at D20 | Day 20
  This outcome evaluates the delay between inclusion and hospitalization at D20.
Effect of treatment on time to hospitalization at D60 | Day 60
  This outcome evaluates the delay between inclusion and hospitalization at D60.
Effect of treatment on Duration of Hospital stay et D20 | Day 20
  This outcome evaluates the duration of patient's Hospital stay at D20.
Effect of treatment on Duration of Hospital stay et D60 | Day 60
  This outcome evaluates the duration of patient's Hospital stay at D60.
Effect of treatment on Duration of symptoms at D20 | Day 20
  This outcome evaluates the duration of symptoms at D20 after treatment.
Effect of treatment on Duration of symptoms at D60 | Day 60
  This outcome evaluates the duration of symptoms at D60 after treatment.
Incidence of Treatment-Emergent Adverse Events | Month 6
  This outcome measures the number of participants with treatment-related adverse events as assessed by CTCAE v4.0, at the end of study.

OTHER OUTCOMES:
Effect of treatment on chest radiological features | Month 6
  This outcome evaluates the chest radiological features on Chest HRCT, at 6 months, after treatment.
Effect of treatment on respiratory capacity | Month 6
  This outcome evaluates the Pulmonary function test at 6 month, after treatment.
Cost consequence analysis | Month 6
  This ouctome eavaluates costs and consequences which will be presented for each stakeholder in a disaggregated way at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Naccache, MD, Principal Investigator — Fondation Hôpital Saint-Joseph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Liang WH, Zhao Y, Liang HR, Chen ZS, Li YM, Liu XQ, Chen RC, Tang CL, Wang T, Ou CQ, Li L, Chen PY, Sang L, Wang W, Li JF, Li CC, Ou LM, Cheng B, Xiong S, Ni ZY, Xiang J, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX; China Medical Treatment Expert Group for COVID-19. Comorbidity and its impact on 1590 patients with COVID-19 in China: a nationwide analysis. Eur Respir J. 2020 May 14;55(5):2000547. doi: 10.1183/13993003.00547-2020. Print 2020 May. PMID 32217650
- [Background] Khan AA, Slifer TR, Araujo FG, Remington JS. Effect of clarithromycin and azithromycin on production of cytokines by human monocytes. Int J Antimicrob Agents. 1999 Feb;11(2):121-32. doi: 10.1016/s0924-8579(98)00091-0. PMID 10221415
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Chan JF, Yao Y, Yeung ML, Deng W, Bao L, Jia L, Li F, Xiao C, Gao H, Yu P, Cai JP, Chu H, Zhou J, Chen H, Qin C, Yuen KY. Treatment With Lopinavir/Ritonavir or Interferon-beta1b Improves Outcome of MERS-CoV Infection in a Nonhuman Primate Model of Common Marmoset. J Infect Dis. 2015 Dec 15;212(12):1904-13. doi: 10.1093/infdis/jiv392. Epub 2015 Jul 21. PMID 26198719
- [Background] Keyaerts E, Vijgen L, Maes P, Neyts J, Van Ranst M. In vitro inhibition of severe acute respiratory syndrome coronavirus by chloroquine. Biochem Biophys Res Commun. 2004 Oct 8;323(1):264-8. doi: 10.1016/j.bbrc.2004.08.085. PMID 15351731
- [Background] Rolain JM, Colson P, Raoult D. Recycling of chloroquine and its hydroxyl analogue to face bacterial, fungal and viral infections in the 21st century. Int J Antimicrob Agents. 2007 Oct;30(4):297-308. doi: 10.1016/j.ijantimicag.2007.05.015. Epub 2007 Jul 16. PMID 17629679
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Nukoolkarn V, Lee VS, Malaisree M, Aruksakulwong O, Hannongbua S. Molecular dynamic simulations analysis of ritonavir and lopinavir as SARS-CoV 3CL(pro) inhibitors. J Theor Biol. 2008 Oct 21;254(4):861-7. doi: 10.1016/j.jtbi.2008.07.030. Epub 2008 Jul 29. PMID 18706430
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Yogasundaram H, Putko BN, Tien J, Paterson DI, Cujec B, Ringrose J, Oudit GY. Hydroxychloroquine-induced cardiomyopathy: case report, pathophysiology, diagnosis, and treatment. Can J Cardiol. 2014 Dec;30(12):1706-15. doi: 10.1016/j.cjca.2014.08.016. Epub 2014 Aug 23. PMID 25475472